CLINICAL TRIAL: NCT00185965
Title: Le23 CPG: A Phase 1-2 Study of Intratumoral Injection of CPG 7909, A TLR 9 Agonist, Combined With Local Radiation in Recurrent Low-Grade Lymphomas
Brief Title: CPG 7909 + Local Radiotherapy in Recurrent Low-Grade Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ronald Levy (Other)
Collaborators: Lymphoma Research Foundation (Other); American Society of Clinical Oncology (Other)
Responsible Party: Sponsor-Investigator, Ronald Levy, Robert K. and Helen K. Summy Professor in the School of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13063; 80057 (Other: Stanford University Alternate IRB Number); LYMNHL0014 (Other: OnCore)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Non-Hodgkin Lymphoma; Mycosis Fungoides
Keywords: non-Hodgkin; lymphoma; mycosis; fungoides
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Mycosis Fungoides; Lymphoma; Mycoses | interventions — ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lymphoma, B-cell low-grade (BCL) (Experimental): Recurrent low-grade B-cell lymphoma patients (at least one prior treatment failure)
  Interventions: Drug: CPG 7909
- Mycosis fungoides (MF) (Experimental): Mycosis fungoides patients must have failed or have been intolerant of at least 1 topical or 1 systemic treatment
  Recurrent mycosis fungoides patients (at least one prior failure of topical or systemic treatment)
  Interventions: Drug: CPG 7909

INTERVENTIONS:
Drug: CPG 7909 — 6 mg intratumoral injection, administered immediately before 2 Gy radiotherapy (RT) to a designated tumor lesion, about 24 hours later after a 2nd 2 Gy RT dose, then weekly for 8 additional weeks (total of 10 injections).
  Other Names: PF-3512676; CPG-enriched TLR9 agonist; CPG

SUMMARY:
Brief summary TBD

DETAILED DESCRIPTION:
This is a single institution phase 1-2 trial to evaluate the safety, feasibility and efficacy of CpG injections (4 intratumoral injections followed by 6 peri-tumoral injections) combined with local irradiation in patients with recurrent low-grade lymphomas.

Patients will receive low-dose radiotherapy to a single tumor site on days 1 and 2 (2 Gy each day). CpG injections will be administered into the same tumor site within the 24 hours before and the 24 hours after the radiation, and on days 8 and 15. Weekly doses of CpG will be then administered subcutaneously in the region of previous injections for 6 additional doses.

ELIGIBILITY:
Inclusion Criteria:Patients must meet all of the following criteria in order to be eligible for entry into the trial.

* Biopsy confirmed low-grade B-cell lymphoma of any initial stage or mycosis fungoides of stage IB-IVA. B-cell lymphoma patients must have failed at least one prior treatment. Mycosis fungoides patients must have failed or have been intolerant of at least 2 topical or one systemic treatment.
* Patients must have at least one site of disease that is accessible for intratumoral injection of CpG percutaneously
* Tumor specimens must be available for immunological studies either from a previous biopsy or a new biopsy obtained before the initiation of the treatment.
* Patients must have measurable disease other than the injection site or biopsy site.
* 18 years of age or older
* Karnofsky Performance Status (KPS) of > 70.
* Adequate bone marrow function: WBC>4,000uL, hemoglobin > 10g/dL; platelet count >100,000/mm3; ANC> 1000.
* Adequate hepatic function: bilirubin <= 1.5 mg/dL; SGOT/SGPT<3xupper limit of normal
* Adequate renal function: serum creatinine <= 2.0mg/dL.
* Required wash out periods for prior therapy:

  * Topical therapy: 2 weeks
  * Chemotherapy: 4 weeks
  * Radiotherapy (including photo therapy): 4 weeks
  * Systemic biological therapy for mycosis fungoides: 4 weeks
  * Other investigational therapy: 4weeks
  * Rituximab: 12 weeks
* Patients of reproductive potential and their partners must agree to use an effective (>90% reliability) form of contraception during the study and for 4 weeks following the last study drug administration.
* Women of reproductive potential must have negative urine pregnancy test.
* Life expectancy greater than 4 months.
* Able to comply with the treatment schedule.

Exclusion Criteria:A patient may not be enrolled in the trial if any of the following criteria are met.

* Pre-existing autoimmune or antibody mediated disease including: systemic lupus, erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, but excluding controlled thyroid disease, or the presence of autoantibodies without clinical autoimmune disease.
* Known history of human immunodeficiency virus (HIV), hepatitis B or hepatitis C (active, prior treatment, or both).
* Patients with active infection or with a fever >38.50 C within three days prior to the first scheduled treatment.
* CNS metastases
* Prior malignancy (active within 5 years of screening) except basal cell or completely excised non-invasive squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix.
* History of allergic reactions attributed to compounds of similar composition to CpG 7909
* Current anticoagulant therapy (ASA<= 325mg/day allowed).
* Significant cardiovascular disease (i.e. NYHA class 3 congestive heart failure; myocardial infarction with the past 6 months; unstable angina; coronary angioplasty with the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
* Pregnant or lactating.
* Any other medical history, including laboratory results, deemed by the investigator to be likely to interfere with their participation in the study, or to interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Levy, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Kim YH, Gratzinger D, Harrison C, Brody JD, Czerwinski DK, Ai WZ, Morales A, Abdulla F, Xing L, Navi D, Tibshirani RJ, Advani RH, Lingala B, Shah S, Hoppe RT, Levy R. In situ vaccination against mycosis fungoides by intratumoral injection of a TLR9 agonist combined with radiation: a phase 1/2 study. Blood. 2012 Jan 12;119(2):355-63. doi: 10.1182/blood-2011-05-355222. Epub 2011 Nov 1. PMID 22045986
- [Result] Brody JD, Ai WZ, Czerwinski DK, Torchia JA, Levy M, Advani RH, Kim YH, Hoppe RT, Knox SJ, Shin LK, Wapnir I, Tibshirani RJ, Levy R. In situ vaccination with a TLR9 agonist induces systemic lymphoma regression: a phase I/II study. J Clin Oncol. 2010 Oct 1;28(28):4324-32. doi: 10.1200/JCO.2010.28.9793. Epub 2010 Aug 9. PMID 20697067

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycosis Fungoides (MF): Recurrent mycosis fungoides patients (at least one prior failure of topical or systemic treatment)
  CPG 7909: 6 mg intratumoral injection, administered immediately before 2 Gy radiotherapy (RT) to a designated tumor lesion, about 24 hours later after a 2nd 2 Gy RT dose, then weekly for 8 additional weeks (total of 10 injections).
Period: Overall Study
Arm/Group | Lymphoma, B-cell Low-grade (BCL) | Mycosis Fungoides (MF)
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lymphoma, B-cell Low-grade (BCL) | Mycosis Fungoides (MF) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Full Range); unit: years] | 62 [38 to 65] | 57 [18 to 71] | 60 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) consisting of Complete Response (CR) + Partial Response (PR), not including Stable Disease (SD)
Time Frame: 12 weeks
Measure: Number; unit: percentage of treated subjects
Arm/Group | Lymphoma, B-cell Low-grade (BCL) | Mycosis Fungoides (MF)
Number analyzed (Participants) | 15 | 14
percentage of treated subjects | 26.7 | 35.7

ADVERSE EVENTS:
Arm/Group | Lymphoma, B-cell Low-grade (BCL) | Mycosis Fungoides (MF)
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 5/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphoma, B-cell Low-grade (BCL) (N=15) | Mycosis Fungoides (MF) (N=15)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphoma, B-cell Low-grade (BCL) (N=15) | Mycosis Fungoides (MF) (N=15)
Flu like symptoms (General disorders) | 5 (5) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 14 (14)
Chills (General disorders) | 0 (0) | 14 (14)
Fatigue (General disorders) | 0 (0) | 13 (13)
Headache (Nervous system disorders) | 0 (0) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (10)
Fever (General disorders) | 0 (0) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palpitation (Cardiac disorders) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No